CLINICAL TRIAL: NCT03214952
Title: Drug Use Surveillance of Takecab Tablets for "Gastric Ulcer, Duodenal Ulcer, and Reflux Esophagitis"
Brief Title: Drug Use Surveillance of Vonoprazan for "Gastric Ulcer, Duodenal Ulcer, and Reflux Esophagitis"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vonoprazan-5001; JapicCTI-163177 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2017-07-09; First posted 2017-07-12 (Actual); Results first posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-11

CONDITIONS: Gastric Ulcer, Duodenal Ulcer, and Reflux Esophagitis
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer; Esophagitis, Peptic | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vonoprazan 20 mg: The usual adult dosage for oral use is 20 mg of vonoprazan administered orally once daily. An 8-week treatment for gastric ulcer and a 6-week treatment for duodenal ulcer. For reflux esophagitis, the usual adult dosage for oral use was administered for a total of 4 weeks of treatment, and if that dosing proved insufficient, the administration may have been extended, but for no longer than 8 weeks of treatment. Participants received vonoprazan as part of a routine medical care.
  Interventions: Drug: Vonoprazan

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan tablets
  Other Names: Takecab tablets; TAK-438

SUMMARY:
The purpose of this survey is to evaluate the safety and effectiveness of vonoprazan tablets in patients with gastric ulcer, duodenal ulcer, and reflux esophagitis in the routine clinical setting.

DETAILED DESCRIPTION:
The drug being tested in this survey is called vonoprazan. Vonoprazan is being tested to treat patients who have gastric ulcer, duodenal ulcer, and reflux esophagitis.

This survey will look at the safety and effectiveness of vonoprazan in patients with gastric ulcer, duodenal ulcer, and reflux esophagitis in the routine clinical setting. The survey will enroll approximately 3000 participants.

- Vonoprazan 20 mg

This multi-center survey will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

- Participants with gastric ulcer, duodenal ulcer, and reflux esophagitis

Exclusion Criteria:

* Participants with previous history of hypersensitivity to ingredients in Takecab tablets
* Participants taking atazanavir sulfate or rilpivirine hydrochloride
* Participants meeting the criteria of scarring stage (S1, S2) of endoscopic classification defined by Sakita and Miwa at the start of the treatment with Takecab tablets, in the case that the target disease is gastric ulcer or duodenal ulcer
* Participants meeting the criteria of Grade N or Grade M of Los Angeles classification (Hoshihara's modification) at the start of the treatment with Takecab tablets, in the case that the target disease is reflux esophagitis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of participants with a diagnosis of gastric ulcer, duodenal ulcer, and reflux esophagitis and receive Vonoprazan in the routine clinical setting.
Sampling Method: Non-Probability Sample
Enrollment: 3183 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 291 investigative sites in Japan, from 01 March 2016 to 31 October 2018.
Pre-assignment Details: Participants with a historical diagnosis of gastric ulcer, duodenal ulcer, and reflux esophagitis were enrolled. Participants received vonoprazan as part of a routine medical care.
Period: Overall Study
Arm/Group | Vonoprazan 20 mg
Started | 3183
Completed | 3125
Not Completed | 58
Not completed — Protocol Deviation | 45
Not completed — Case Report Forms Uncollected | 13

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Vonoprazan 20 mg
Number analyzed (Participants) | 3125
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (16.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1375
  Male | 1750
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 3125
Target Conditions of Study Treatment [Count of Participants; unit: Participants] — Participants could be counted in more than one category, including duplicates.
  Participants
    Gastric Ulcer | 1097
    Duodenal Ulcer | 578
    Reflux Esophagitis | 1540
Duration of Diagnosis of Gastric Ulcer, Duodenal Ulcer, and Reflux Esophagitis [Mean (Standard Deviation); unit: Days] — Mean duration between first time of diagnosis of gastric ulcer, duodenal ulcer, and reflux esophagitis and start of survey was reported. Population: The number analyzed is the number of participants with data available for analysis.
  Days
    number analyzed (Participants) | 3045
    (all) | 38.3 (281.47)
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient and inpatient.
  Participants
    Outpatient | 2744
    Inpatient | 381
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — Number of participants who had or did not have a liability or tendency to suffer from hypersensitivity was reported.
  Participants
    Had No Predisposition to Hypersensitivity | 2893
    Had Predisposition to Hypersensitivity | 117
    Unknown | 115
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Medical Complications | 1652
    Had Medical Complications | 1473
Medical History of Gastric Ulcer, Duodenal Ulcer, and Reflux Esophagitis [Count of Participants; unit: Participants] — Number of participants with or without medical history of gastric ulcer, duodenal ulcer, and reflux esophagitis was reported.
  Participants
    Had No Medical History | 2256
    Had Medical History | 590
    Unknown | 279
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  Centimeters (cm)
    number analyzed (Participants) | 1770
    (all) | 161.01 (10.142)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 1830
    (all) | 60.46 (13.377)
BMI [Mean (Standard Deviation); unit: Kilogram (kg)/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  Kilogram (kg)/meter (m)^2
    number analyzed (Participants) | 1757
    (all) | 23.15 (3.798)
Helicobacter Pylori Infection [Count of Participants; unit: Participants] — Number of participants with or without history of H. pylori infection was reported. "Negative" indicates the absence of H. pylori infection, "Positive" indicates presence of the infection.
  Participants
    Negative | 1492
    Positive | 862
    Unknown | 771
Medical History of Esophageal Hiatal Hernia [Count of Participants; unit: Participants] — Number of participants with or without medical history of esophageal hiatal hernia was reported.
  Participants
    Had No Esophageal Hiatal Hernia | 1920
    Had Esophageal Hiatal Hernia | 1034
    Unknown | 171
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 1258
  Current Smoker | 626
  Ex-Smoker | 429
  Unknown | 812
Drinking Habits [Count of Participants; unit: Participants] — Participants who answered Yes or No for a question "Drink Alcohol Almost Every Day?" were reported.
  Participants
    Yes | 784
    No | 1704
    Unknown | 637
Endoscopic Findings; Gastric Ulcer [Count of Participants; unit: Participants] — Endoscopic findings of ulcer were classified per Sakita-Miwa Classification as follows; Active stage: A1 and A2, Healing stage: H1 and H2, Scarring stage: S1 and S2. Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 1031
    Active stage, A1 and A2 | 784
    Healing stage, H1 and H2 | 247
Endoscopic Findings; Duodenal Ulcer [Count of Participants; unit: Participants] — Endoscopic findings of ulcer were classified per Sakita-Miwa Classification as follows; Active stage: A1 and A2, Healing stage: H1 and H2, Scarring stage: S1 and S2. Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 535
    Active stage, A1 and A2 | 370
    Healing stage, H1 and H2 | 165
Endoscopic Findings; Reflux Esophagitis [Count of Participants; unit: Participants] — Endoscopic findings were assessed using the modified Los Angeles (LA) classification. The modified LA classification graded as follows- Grade N: normal mucosa; Grade M: minimal changes to the mucosa, such as erythema and/or whitish turbidity; Grade A: non-confluent mucosal breaks less than (<) 5 mm in length; Grade B: nonconfluent mucosal breaks greater than or equal to (>=) 5mm in length; Grade C: confluent mucosal breaks <75% circumferential; Grade D: confluent mucosal breaks greater than (>) 75% circumferential. Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 1276
    Grade A | 626
    Grade B | 389
    Grade C | 171
    Grade D | 90
Prior Treatment for Gastric Ulcer, Duodenal Ulcer, and Reflux Esophagitis [Count of Participants; unit: Participants] — Number of participants who had or had not been treated for gastric ulcer, duodenal ulcer, and reflux esophagitis was reported.
  Participants
    Had No Prior Treatment | 2280
    Had Prior Treatment | 791
    Unknown | 54
Duration of Prior Treatment [Count of Participants; unit: Participants] — Duration of prior treatment for gastric ulcer, duodenal ulcer, and reflux esophagitis was categorized as < 1 month, >= 1 month and < 2 months, and >= 2 months by number of participants. Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 791
    < 1 month | 436
    >= 1 month and < 2 months | 56
    >= 2 months | 299

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Gastric Ulcer Who Had One or More Adverse Drug Reactions
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction refers to AE related to the administered drug.
Time Frame: Up to 8 weeks
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey. Participants who treated for gastric ulcer within the Safety Analysis Set were analyzed for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vonoprazan 20 mg
Number analyzed (Participants) | 1097
Percentage of Participants | 1.00

2. Primary Outcome: Percentage of Participants With Duodenal Ulcer Who Had One or More Adverse Drug Reactions
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction refers to AE related to the administered drug.
Time Frame: Up to 6 weeks
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey. Participants who treated for duodenal ulcer within the Safety Analysis Set were analyzed for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vonoprazan 20 mg
Number analyzed (Participants) | 578
Percentage of Participants | 1.21

3. Primary Outcome: Percentage of Participants With Reflux Esophagitis Who Had One or More Adverse Drug Reactions
Description: as for outcome 2
Time Frame: Up to 8 weeks
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey. Participants who treated for reflux esophagitis within the Safety Analysis Set were analyzed for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vonoprazan 20 mg
Number analyzed (Participants) | 1540
Percentage of Participants | 0.78

4. Secondary Outcome: Endoscopic Cure Rate in Participants With Gastric Ulcer
Description: Endoscopic cure rate was defined as a percentage of participants treated for gastric ulcer who classified as Scarring stage at the end of survey per Sakita-Miwa Classification. Endoscopic findings of ulcer were classified per Sakita-Miwa Classification as follows; Active stage: A1 and A2, Healing stage: H1 and H2, Scarring stage: S1 and S2.
Time Frame: Up to 8 weeks
Population: Efficacy assessment population, participants who completed the survey and evaluable for efficacy; Participants who treated for gastric ulcer within Efficacy assessment population and evaluable for endoscopic cure rate were analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vonoprazan 20 mg
Number analyzed (Participants) | 484
Percentage of Participants | 78.72 [74.80 to 82.28]

5. Secondary Outcome: Endoscopic Cure Rate in Participants With Duodenal Ulcer
Description: Endoscopic cure rate was defined as a percentage of participants treated for duodenal ulcer who classified as Scarring stage at the end of survey per Sakita-Miwa Classification. Endoscopic findings of ulcer were classified per Sakita-Miwa Classification as follows; Active stage: A1 and A2, Healing stage: H1 and H2, Scarring stage: S1 and S2.
Time Frame: Up to 6 weeks
Population: Efficacy assessment population, participants who completed the survey and evaluable for efficacy; Participants who treated for duodenal ulcer within Efficacy assessment population and evaluable for endoscopic cure rate were analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vonoprazan 20 mg
Number analyzed (Participants) | 234
Percentage of Participants | 88.46 [83.66 to 92.26]

6. Secondary Outcome: Endoscopic Cure Rate in Participants With Reflux Esophagitis
Description: Endoscopic cure rate was defined as a percentage of participants who treated for reflux esophagitis and met the criteria of Grade N or M in the modified Los Angeles (LA) classification at the end of survey. Grade N: normal mucosa; Grade M: minimal changes to the mucosa, such as erythema and/or whitish turbidity.
Time Frame: Up to 8 weeks
Population: Efficacy assessment population, participants who completed the survey and evaluable for efficacy; Participants who treated for reflux esophagitis within Efficacy assessment population and evaluable for endoscopic cure rate were analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vonoprazan 20 mg
Number analyzed (Participants) | 226
Percentage of Participants | 65.04 [58.44 to 71.25]

7. Secondary Outcome: Percentage of Participants With Gastric Ulcer Whose Subjective Symptoms Improved
Description: Percentage of participants who treated for gastric ulcer and whose subjective symptoms, including heartburn, acid reflux, postprandial fullness, early satiation, epigastric pain, epigastric burning, abdominal bloating, nausea/vomiting, belching and anorexia, were improved was reported. Presence or absence and severity of subjective symptoms were graded as asymptomatic, mild (occasionally or slightly symptomatic), moderate (considerably symptomatic), and severe (unendurably symptomatic). Participants with whose subjective symptom was improved by one grade or better were defined as "Improved".
Time Frame: Baseline and at the end of the survey (up to 8 weeks)
Population: Efficacy assessment population, participants who completed the survey and evaluable for efficacy; Participants who treated for gastric ulcer within Efficacy assessment population and evaluable for subjective symptoms were analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vonoprazan 20 mg
Number analyzed (Participants) | 1060
Percentage of Participants
  Heartburn: number analyzed (Participants) | 211
  Heartburn | 96.68 [93.28 to 98.66]
  Acid Reflux: number analyzed (Participants) | 159
  Acid Reflux | 96.86 [92.81 to 98.97]
  Postprandial Fullness: number analyzed (Participants) | 307
  Postprandial Fullness | 96.09 [93.27 to 97.96]
  Early Satiation: number analyzed (Participants) | 171
  Early Satiation | 97.08 [93.31 to 99.04]
  Epigastric Pain: number analyzed (Participants) | 654
  Epigastric Pain | 98.78 [97.60 to 99.47]
  Epigastric Burning: number analyzed (Participants) | 168
  Epigastric Burning | 97.62 [94.02 to 99.35]
  Abdominal Bloating: number analyzed (Participants) | 207
  Abdominal Bloating | 95.65 [91.91 to 97.99]
  Nausea/Vomiting: number analyzed (Participants) | 242
  Nausea/Vomiting | 97.52 [94.68 to 99.08]
  Belching: number analyzed (Participants) | 120
  Belching | 91.67 [85.21 to 95.93]
  Anorexia: number analyzed (Participants) | 337
  Anorexia | 98.22 [96.17 to 99.34]

8. Secondary Outcome: Percentage of Participants With Duodenal Ulcer Whose Subjective Symptoms Improved
Description: Percentage of participants who treated for duodenal ulcer and whose subjective symptoms, including heartburn, acid reflux, postprandial fullness, early satiation, epigastric pain, epigastric burning, abdominal bloating, nausea/vomiting, belching and anorexia, were improved was reported. Presence or absence and severity of subjective symptoms were graded as asymptomatic, mild (occasionally or slightly symptomatic), moderate (considerably symptomatic), and severe (unendurably symptomatic). Participants with whose subjective symptom was improved by one grade or better were defined as "Improved".
Time Frame: Baseline and at the end of the survey (up to 6 weeks)
Population: Efficacy assessment population, participants who completed the survey and evaluable for efficacy; Participants who treated for duodenal ulcer within Efficacy assessment population and evaluable for subjective symptoms were analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vonoprazan 20 mg
Number analyzed (Participants) | 577
Percentage of Participants
  Heartburn: number analyzed (Participants) | 98
  Heartburn | 96.94 [91.31 to 99.36]
  Acid Reflux: number analyzed (Participants) | 72
  Acid Reflux | 97.22 [90.32 to 99.66]
  Postprandial Fullness: number analyzed (Participants) | 138
  Postprandial Fullness | 95.65 [90.78 to 98.39]
  Early Satiation: number analyzed (Participants) | 82
  Early Satiation | 98.78 [93.39 to 99.97]
  Epigastric Pain: number analyzed (Participants) | 351
  Epigastric Pain | 98.58 [96.71 to 99.54]
  Epigastric Burning: number analyzed (Participants) | 67
  Epigastric Burning | 100.00 [94.64 to 100.00]
  Abdominal Bloating: number analyzed (Participants) | 97
  Abdominal Bloating | 93.81 [87.02 to 97.70]
  Nausea/Vomiting: number analyzed (Participants) | 130
  Nausea/Vomiting | 96.92 [92.31 to 99.16]
  Belching: number analyzed (Participants) | 62
  Belching | 93.55 [84.30 to 98.21]
  Anorexia: number analyzed (Participants) | 143
  Anorexia | 99.30 [96.17 to 99.98]

9. Secondary Outcome: Percentage of Participants With Reflux Esophagitis Whose Subjective Symptoms Improved
Description: Percentage of participants who treated for reflux esophagitis and whose subjective symptoms, including heartburn, acid reflux, postprandial fullness, early satiation, epigastric pain, epigastric burning, abdominal bloating, nausea/vomiting, belching and anorexia, were improved was reported. Presence or absence and severity of subjective symptoms were graded as asymptomatic, mild (occasionally or slightly symptomatic), moderate (considerably symptomatic), and severe (unendurably symptomatic). Participants with whose subjective symptom was improved by one grade or better were defined as "Improved".
Time Frame: Baseline and at the end of the survey (up to 8 weeks)
Population: Efficacy assessment population, participants who completed the survey and evaluable for efficacy; Participants who treated for reflux esophagitis within Efficacy assessment population and evaluable for subjective symptoms were analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vonoprazan 20 mg
Number analyzed (Participants) | 1527
Percentage of Participants
  Heartburn: number analyzed (Participants) | 1027
  Heartburn | 96.20 [94.85 to 97.29]
  Acid Reflux: number analyzed (Participants) | 776
  Acid Reflux | 94.33 [92.46 to 95.85]
  Postprandial Fullness: number analyzed (Participants) | 546
  Postprandial Fullness | 93.22 [90.78 to 95.18]
  Early Satiation: number analyzed (Participants) | 236
  Early Satiation | 92.37 [88.21 to 95.42]
  Epigastric Pain: number analyzed (Participants) | 522
  Epigastric Pain | 95.79 [93.69 to 97.34]
  Epigastric Burning: number analyzed (Participants) | 396
  Epigastric Burning | 96.72 [94.45 to 98.24]
  Abdominal Bloating: number analyzed (Participants) | 281
  Abdominal Bloating | 90.04 [85.92 to 93.28]
  Nausea/Vomiting: number analyzed (Participants) | 265
  Nausea/Vomiting | 95.47 [92.22 to 97.64]
  Belching: number analyzed (Participants) | 405
  Belching | 89.38 [85.97 to 92.21]
  Anorexia: number analyzed (Participants) | 265
  Anorexia | 93.96 [90.38 to 96.51]

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Vonoprazan 20 mg
All-Cause Mortality (participants affected / at risk) | 6/3125
Serious Adverse Events (participants affected / at risk) | 20/3125
Other Adverse Events (participants affected / at risk) | 10/3125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 20 mg (N=3125)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Alcoholic psychosis (Psychiatric disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Aortic aneurysm rupture (Vascular disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Pyrexia (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 20 mg (N=3125)
Nausea (Gastrointestinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT03214952/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT03214952/SAP_001.pdf